CLINICAL TRIAL: NCT00025883
Title: Long-Term Efficacy of Leptin Replacement in Treatment of Lipodystrophy
Brief Title: Leptin to Treat Lipodystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020022; 02-DK-0022 (Other: National Institutes of Health Clinical Center)
Record Dates: First submitted 2001-10-27; First posted 2001-10-29 (Estimated); Results first posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Lipodystrophy
Keywords: Lipoatrophic Diabetes; Diabetes Mellitus; Hypertriglyceridemia; NASH; Lipodystrophy; Leptin; Diabetes
MeSH Terms: conditions — Lipodystrophy; Diabetes Mellitus, Lipoatrophic; Diabetes Mellitus; Hypertriglyceridemia | interventions — metreleptin; Leptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metreleptin (Experimental): subcutaneous metreleptin injections in one to two daily doses ranging from 0.06 to 0.24 mg/kg per day.
  Interventions: Drug: Metreleptin

INTERVENTIONS:
Drug: Metreleptin — Drug treatment
  Other Names: Leptin

SUMMARY:
This study will evaluate the safety and effectiveness of leptin replacement therapy in patients with lipodystrophy (also called lipoatrophy). Patients have a total or partial loss of fat cells. They also lack the hormone leptin, which is produced by fat cells. The leptin deficiency usually causes high blood lipid (fat) levels and insulin resistance that may lead to diabetes. Patients may have hormone imbalances, fertility problems, large appetite, and liver disease due to fat accumulation.

Patients age greater than or equal to 6 months with significant lipodystrophy may be eligible for this study. Participants will be admitted to the NIH Clinical Center for 10 days for the following studies before beginning 12 months of leptin therapy:

* Insulin tolerance test
* Ultrasound of the liver and, if abnormalities are found, possibly liver biopsies.
* Fasting blood tests
* Resting metabolic rate
* Magnetic resonance imaging of the liver and other organs, and of muscle and fat.
* Pelvic ultrasound in women to detect ovarian cysts.
* Estimation of body fat
* Oral glucose tolerance test
* Intravenous glucose tolerance test
* Appetite level and food intake
* Hormone function tests
* Questionnaires to assess activity and mood
* 24-hour urine collections

Additional studies may include blood tests for genetic studies of lipodystrophy, a muscle biopsy to study muscle proteins involved in regulating energy expenditure before and after leptin replacement, and examination of a surgical specimen (if available) to study molecules that may be involved in energy storage and use.

When the above tests are completed, leptin therapy begins. The drug is injected under the skin twice a day for 4 months and then once a day, if feasible. The dose is increased at the 1- and 2-month visits. Follow-up visits at 1, 2, 4, 6, 8 and 12 months after therapy starts include a physical examination, blood tests and a meeting with a dietitian. At the end of 12 months, all baseline studies described above are repeated. Patients record their symptoms weekly throughout the study. Those with diabetes measure their blood glucose levels daily before each meal and at bedtime.

DETAILED DESCRIPTION:
Lipoatrophic diabetes is a syndrome characterized by insulin resistance in association with a paucity of adipose tissue. Patients with severe lipoatrophy die prematurely, typically from the complications of diabetes or liver disease. Experiments with lipoatrophic mice suggest that the insulin resistance is caused by the lack of adipose tissue. Adipose tissue normally produces leptin, a hormone that increases insulin action. For the last fourteen years, we have been studying the extent to which leptin deficiency causes diabetes in lipoatrophic patients. In fact, in our initial study we have seen nearly 60% amelioration of fasting glucose, triglycerides and free fatty acid levels and about 2% actual decreases from baseline HbA1c levels with 4 months of leptin replacement therapy. This response has continued to be sustained, as we continue to follow patients that have now received leptin replacement therapy for fourteen years.

This is an open-labeled study. The study monitors the safety and efficacy of recombinant methionyl human leptin (A-100) replacement in children and adults. We are looking at the long-term effects of leptin replacement on extended therapy. In this long-term replacement protocol, we will monitor metabolic control (e.g. glucose, insulin, and triglyceride levels) as primary outcome measures. Ancillary studies will evaluate the effect of Metreleptin on other hormonal axes, growth and development and on liver pathology.

We continue to evaluate the efficacy in a broader leptin deficient population of patients with lipodystrophy. Current inclusion criteria in patients greater than or equal to 5 years include female patients with leptin levels < 12 ng/mL and male patients with leptin levels < 8 ng/mL. We continue to seek patients who meet these criteria. In children ages 6 months 5 years, we will use a cut-off leptin level of 6 ng/mL in both genders.

Patients who are greater than or equal to age 5 years will be evaluated every 6 months during the first year of therapy. If no improvements are seen after 6 months of therapy, then the study medication may be increased to 150% of the predicted dose (0.09mg/kg/day for males and girls less than 10 years of age/ 0.12mg/kg/day for females 10 years of age and older) from 6 months to 1 year on therapy. If no improvements are seen after increasing to 150% of the predicted dose, then the study medication will be withdrawn. If the patient shows improvements in his/her metabolic parameters while on leptin, the patient will be invited to continue taking the study medication. The investigators will strive for all patients responding to leptin to bring their metabolic parameters into the normal range. The maximum dose of leptin that will be given is 0.24 mg/kg/day for females 10 and older, and 0.12 mg/kg/day for males and females less than 10 years of age. After the first year of treatment, the patient will be evaluated every 6 months through the second year of treatment, and then the study period will end. After two years of treatment, extending the treatment period on an annual basis will be the decision of the patient, principal investigator and Bristol-Myers Squibb (BMS)/AstraZeneca Pharmaceuticals (AZ). Leptin is supplied by BMS/AZ, and is currently only available through research studies. Neither the NIH nor BMS/AZ can guarantee that leptin will be available indefinitely and/or after the study ends. However, leptin was recently approved by the FDA on February 25, 2014, for use in patients with generalized lipodystrophy.

All patient referrals for acceptance into the protocol, are initiated by the physician/health care provider.

ELIGIBILITY:
* INCLUSION CRITERIA:

All ethnic groups.

Males and females.

* Age greater than or equal to 6 months.
* Clinically significant lipodystrophy, identified by the study physician during the physical examination as an absence of fat outside the range of normal variation and/or identified as a disfiguring factor by the patient.

Circulating leptin levels less than 12.0 ng/ml in females and less than 8.0 ng/ml in males as measured by Linco assay on a specimen obtained after an overnight fast. In children ages 6 months 5 years, a circulating leptin level of less than 6 ng/mL will be used. Leptin samples will be run through Millipore Laboratories, who use the Linco Assay, which has been the assay previously used to measure leptin levels throughout this study period.

Presence of at least one of the following metabolic abnormalities:

1. Presence of diabetes as defined by the 2007 ADA criteria

   1. Fasting plasma glucose greater than or equal to 126 mg/dL, or
   2. 2 hour plasma glucose greater than or equal to 200 mg/dL following a 75 gram (1.75gm/kg) oral glucose load, or
   3. Diabetic symptoms with a random plasma glucose greater than or equal to 200 mg/dl
2. Fasting insulin greater than 30 micro units/ml.
3. Fasting hypertriglyceridemia greater than 200 mg/dL or postprandially elevated triglycerides greater than 500 mg/dL when fasting is clinically not indicated (e.g. in infants)

   -Persons with impaired decision-making capacity and who may be unable to provide informed consent may participate in this study per the discretion of the Principal Investigator.

   EXCLUSION CRITERIA:

   Pregnant women, women in their reproductive years who do not use an effective method of birth control, and women currently nursing or lactating within 6 weeks of having completed nursing.

   Exclusions for underlying diseases likely to increase side effects or hinder objective data collection:
   * Known infectious liver disease
   * Known HIV infection
   * Current alcohol or substance abuse
   * Psychiatric disorder impeding competence or compliance
   * Active tuberculosis
   * Use of anorexiogenic drugs
   * Other condition(s) which in the opinion of the clinical investigators would impede completion of the study
   * Subjects who have known hypersensitivity to E. Coli derived proteins.
   * Subjects with acquired lipodystrophy and a hematologic abnormality such as neutropenia and/or lymphadenopathy

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2001-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Gorden, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Burant CF, Sreenan S, Hirano K, Tai TA, Lohmiller J, Lukens J, Davidson NO, Ross S, Graves RA. Troglitazone action is independent of adipose tissue. J Clin Invest. 1997 Dec 1;100(11):2900-8. doi: 10.1172/JCI119839. PMID 9389757
- [Background] Moitra J, Mason MM, Olive M, Krylov D, Gavrilova O, Marcus-Samuels B, Feigenbaum L, Lee E, Aoyama T, Eckhaus M, Reitman ML, Vinson C. Life without white fat: a transgenic mouse. Genes Dev. 1998 Oct 15;12(20):3168-81. doi: 10.1101/gad.12.20.3168. PMID 9784492
- [Background] Cao H, Hegele RA. Nuclear lamin A/C R482Q mutation in canadian kindreds with Dunnigan-type familial partial lipodystrophy. Hum Mol Genet. 2000 Jan 1;9(1):109-12. doi: 10.1093/hmg/9.1.109. PMID 10587585
- [Derived] Okawa MC, Tuska RM, Lightbourne M, Abel BS, Walter M, Dai Y, Cochran E, Brown RJ. Insulin Signaling Through the Insulin Receptor Increases Linear Growth Through Effects on Bone and the GH-IGF-1 Axis. J Clin Endocrinol Metab. 2023 Dec 21;109(1):e96-e106. doi: 10.1210/clinem/dgad491. PMID 37595266
- [Derived] Meral R, Malandrino N, Walter M, Neidert AH, Muniyappa R, Oral EA, Brown RJ. Endogenous Leptin Concentrations Poorly Predict Metreleptin Response in Patients With Partial Lipodystrophy. J Clin Endocrinol Metab. 2022 Mar 24;107(4):e1739-e1751. doi: 10.1210/clinem/dgab760. PMID 34677608
- [Derived] Nguyen ML, Sachdev V, Burklow TR, Li W, Startzell M, Auh S, Brown RJ. Leptin Attenuates Cardiac Hypertrophy in Patients With Generalized Lipodystrophy. J Clin Endocrinol Metab. 2021 Oct 21;106(11):e4327-e4339. doi: 10.1210/clinem/dgab499. PMID 34223895
- [Derived] Sekizkardes H, Cochran E, Malandrino N, Garg A, Brown RJ. Efficacy of Metreleptin Treatment in Familial Partial Lipodystrophy Due to PPARG vs LMNA Pathogenic Variants. J Clin Endocrinol Metab. 2019 Aug 1;104(8):3068-3076. doi: 10.1210/jc.2018-02787. PMID 31194872
- [Derived] Brown RJ, Meehan CA, Cochran E, Rother KI, Kleiner DE, Walter M, Gorden P. Effects of Metreleptin in Pediatric Patients With Lipodystrophy. J Clin Endocrinol Metab. 2017 May 1;102(5):1511-1519. doi: 10.1210/jc.2016-3628. PMID 28324110
- [Derived] Kassai A, Muniyappa R, Levenson AE, Walter MF, Abel BS, Ring M, Taylor SI, Biddinger SB, Skarulis MC, Gorden P, Brown RJ. Effect of Leptin Administration on Circulating Apolipoprotein CIII levels in Patients With Lipodystrophy. J Clin Endocrinol Metab. 2016 Apr;101(4):1790-7. doi: 10.1210/jc.2015-3891. Epub 2016 Feb 22. PMID 26900642
- [Derived] Chan JL, Koda J, Heilig JS, Cochran EK, Gorden P, Oral EA, Brown RJ. Immunogenicity associated with metreleptin treatment in patients with obesity or lipodystrophy. Clin Endocrinol (Oxf). 2016 Jul;85(1):137-49. doi: 10.1111/cen.12980. Epub 2016 Feb 2. PMID 26589105
- [Derived] Diker-Cohen T, Cochran E, Gorden P, Brown RJ. Partial and generalized lipodystrophy: comparison of baseline characteristics and response to metreleptin. J Clin Endocrinol Metab. 2015 May;100(5):1802-10. doi: 10.1210/jc.2014-4491. Epub 2015 Mar 3. PMID 25734254
- [Derived] Christensen JD, Lungu AO, Cochran E, Collins MT, Gafni RI, Reynolds JC, Rother KI, Gorden P, Brown RJ. Bone mineral content in patients with congenital generalized lipodystrophy is unaffected by metreleptin replacement therapy. J Clin Endocrinol Metab. 2014 Aug;99(8):E1493-500. doi: 10.1210/jc.2014-1353. Epub 2014 Jul 29. PMID 25070319
- [Derived] Joseph J, Shamburek RD, Cochran EK, Gorden P, Brown RJ. Lipid regulation in lipodystrophy versus the obesity-associated metabolic syndrome: the dissociation of HDL-C and triglycerides. J Clin Endocrinol Metab. 2014 Sep;99(9):E1676-80. doi: 10.1210/jc.2014-1878. Epub 2014 Jun 13. PMID 24926953
- [Derived] Kamran F, Rother KI, Cochran E, Safar Zadeh E, Gorden P, Brown RJ. Consequences of stopping and restarting leptin in an adolescent with lipodystrophy. Horm Res Paediatr. 2012;78(5-6):320-5. doi: 10.1159/000341398. Epub 2012 Sep 4. PMID 22965160
- [Derived] Chan JL, Lutz K, Cochran E, Huang W, Peters Y, Weyer C, Gorden P. Clinical effects of long-term metreleptin treatment in patients with lipodystrophy. Endocr Pract. 2011 Nov-Dec;17(6):922-32. doi: 10.4158/EP11229.OR. PMID 22068254
- [Derived] Chong AY, Lupsa BC, Cochran EK, Gorden P. Efficacy of leptin therapy in the different forms of human lipodystrophy. Diabetologia. 2010 Jan;53(1):27-35. doi: 10.1007/s00125-009-1502-9. Epub 2009 Sep 2. PMID 19727665
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-DK-0022.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Metreleptin: subcutaneous metreleptin injections in one to two daily doses ranging from 0.06 to 0.24 mg/kg/day.
Period: Overall Study
Arm/Group | Metreleptin
Started | 103
Generalized Lipodystrophy | 63
Partial Lipodystrophy | 40
Completed | 86
Not Completed | 17
Not completed — had atypical progeriod lipodystrophy | 4
Not completed — no baseline data | 1
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — didn't reach 6 months of Metreleptin | 10

BASELINE CHARACTERISTICS:
Groups:
- Metreleptin With Generalized Lipodystrophy: patients with generalized lipodystrophy with subcutaneous metreleptin injection (0.06-0.24 mg/kg/day)
- Metreleptin With Patial Lipodystrophy: patients with partial lipodystrophy with subcutaneous metreleptin injection (0.06-0.24 mg/kg/day)
- Total: Total of all reporting groups
Arm/Group | Metreleptin With Generalized Lipodystrophy | Metreleptin With Patial Lipodystrophy | Total
Number analyzed (Participants) | 55 | 31 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 18 (12) | 35 (14) | 24 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 31 | 73
  Male | 13 | 0 | 13
Pediatric patients [Number; unit: participants]
  aged <20 years | 42 | 7 | 49
  aged >=20 years | 13 | 24 | 37
Body mass index-standard deviation score (BMI-SDS) [Mean (Standard Deviation); unit: units on a scale] — Body mass index -standard deviation score (BMI-SDS) represents a measure of weight, adjusted for height, sex, and age. sample range of BMI-SDS is (-3.23, 1.91). Higher value indicates more body fat.
  units on a scale | 0.26 (0.98) | 0.66 (0.7) | 0.41 (0.9)
Percentage body fat [Mean (Standard Deviation); unit: percentage of body fat] — percentage of body fat
  percentage of body fat | 9 (2) | 22 (4) | 15 (7)
Leptin [Mean (Standard Deviation); unit: ng/mL] | 1.13 (0.74) | 6.23 (3.96) | 3.03 (3.44)
Glucose [Mean (Standard Deviation); unit: mg/dL] | 180 (80) | 182 (87) | 181 (83)
HbA1c [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 8.4 (2.3) | 8.1 (2.2) | 8.3 (2.3)
Fasting insulin [Mean (Standard Deviation); unit: µU/mL] | 122 (318) | 82 (157) | 108 (273)
C-peptide [Mean (Standard Deviation); unit: ng/mL] | 5.61 (4.03) | 3.56 (2.27) | 4.82 (3.62)
Antidiabetic medications per patient [Mean (Standard Deviation); unit: antidiabetic medications] | 1.13 (0.7) | 1.79 (0.68) | 1.36 (0.81)
Insulin users [Number; unit: participants]
  Yes | 30 | 15 | 45
  No | 24 | 14 | 38
  not known | 1 | 2 | 3
Lipid-lowering medications per patient [Mean (Standard Deviation); unit: lipid-lowering medications] | 0.61 (0.84) | 1.07 (1.04) | 0.82 (0.93)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 214 (110) | 235 (147) | 222 (126)
Triglycerides [Geometric Mean (Inter-Quartile Range); unit: mg/dL] | 467 [200 to 847] | 483 [232 to 856] | 473 [200 to 898]
HDL-C [Mean (Standard Deviation); unit: mg/dL] — high-density lipoprotein cholesterol
  mg/dL | 29 (9) | 31 (9) | 30 (9)
LDL-C [Mean (Standard Deviation); unit: mg/dL] — low-density lipoprotein cholesterol
  mg/dL | 104 (50) | 101 (36) | 103 (46)
Vitamin A [Mean (Standard Deviation); unit: µg/dL] | 57 (33) | 73 (20) | 61 (25)
Vitamin E [Mean (Standard Deviation); unit: mg/dL] | 26 (32) | 34 (21) | 31 (28)
25-Hydroxyvitamin D [Mean (Standard Deviation); unit: ng/mL] | 16 (11) | 23 (13) | 19 (12)
PT [Mean (Standard Deviation); unit: sec] — prothrombin time
  sec | 14.2 (1.2) | 13.2 (0.6) | 13.8 (1.1)
International Normalized Ratio (INR) [Mean (Standard Deviation); unit: ratio] | 1.10 (0.14) | 0.98 (0.06) | 1.05 (0.13)
Daily total insulin units per patient [Mean (Standard Deviation); unit: insulin units] | 625 (1099) | 278 (214) | 362 (620)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Glycosylated Hemoglobin at Baseline, 6 Months, and 12 Months on Treatment With Metreleptin
Description: Percentage of glycosylated hemoglobin at Baseline, 6 months, and 12 months on treatment with metreleptin
Time Frame: Baseline, 6 months, 12 months
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Groups:
- Generalized Lipodystrophy (GLD): patients with generalized lipodystrophy (GLD) with initiation of subcutaneous metreleptin injection (0.06-0.24 mg/kg/day)
- Partial Lipodystrophy (PLD): patients with partial lipodystrophy (PLD) with initiation of subcutaneous metreleptin injection (0.06-0.24 mg/kg/day)
Arm/Group | Generalized Lipodystrophy (GLD) | Partial Lipodystrophy (PLD)
Number analyzed (Participants) | 55 | 31
percentage of glycated hemoglobin
  Baseline | 8.4 (2.3) | 8.1 (2.2)
  6 months | 6.6 (1.7) | 7.2 (1.2)
  12 months | 6.4 (1.5) | 7.3 (1.6)
Statistical Analysis 1: Comparison: Generalized Lipodystrophy (GLD); A null hypothesis of interest is there is no significant change over three time points (baseline, 6 months, 12 months) in response to metreleptin within GLD group; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Partial Lipodystrophy (PLD); A null hypothesis of interest is there is no significant change over three time points (baseline, 6 months, 12 months) in response to metreleptin within PLD group; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis

2. Primary Outcome: Triglycerides at Baseline, 6 Months, and 12 Months on Treatment With Metreleptin
Time Frame: Baseline, 6 months, 12 months
Measure: Geometric Mean (Inter-Quartile Range); unit: mg/dL
Arm/Group | Generalized Lipodystrophy (GLD) | Partial Lipodystrophy (PLD)
Number analyzed (Participants) | 55 | 31
mg/dL
  Baseline | 467 [200 to 847] | 483 [232 to 856]
  6 months | 198 [122 to 283] | 339 [211 to 530]
  12 months | 180 [106 to 312] | 326 [175 to 478]
Statistical Analysis 1: Comparison: Generalized Lipodystrophy (GLD); Triglycerides were log transformed for analysis due to non-normal distribution. Changes in triglycedies in response to metreleptin over three time points (baseline, 6 months, 12 months) are tested within GLD group; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: Partial Lipodystrophy (PLD); Triglycerides were log transformed for analysis due to non-normal distribution. Changes in triglycedies in response to metreleptin over three time points (baseline, 6 months, 12 months) are tested within PLD group; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Metreleptin: subcutaneous metreleptin injection (0.06-0.24 mg/kg/day)
Arm/Group | Metreleptin
Serious Adverse Events (participants affected / at risk) | 10/103
Other Adverse Events (participants affected / at risk) | 64/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metreleptin (N=103)
Abdominal pain requiring hospitalization (Gastrointestinal disorders) | 1 (5)
Acute exacerbation of pancreatitis (Gastrointestinal disorders) | 1 (1)
Severe acute bronchitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Osteomyelitis (Gastrointestinal disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2)
Group B streptococcus bacteremia (Infections and infestations) | 1 (1)
Exacerbations of heart failure (Cardiac disorders) | 2 (5)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Ovarian cyst requiring bilateral oophorectomy and total abdominal hysterectomy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metreleptin (N=103)
Abdominal pain (Gastrointestinal disorders) | 8 (9)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15 (19)
Infection (Infections and infestations) | 7 (12)
Anxiety (General disorders) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Hypoglycemia (Endocrine disorders) | 10 (12)
Weight loss (Metabolism and nutrition disorders) | 12 (12)
tumor, benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Fatigue (Endocrine disorders) | 7 (8)
Insomnia (General disorders) | 5 (5)
Headache (General disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 9 (9)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Decreased appetite (Gastrointestinal disorders) | 4 (4)
Joins pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Depression (General disorders) | 4 (4)
Iron deficiency (Blood and lymphatic system disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes